CLINICAL TRIAL: NCT04471168
Title: Interest of Auriculotherapy in the Management of Chronic Insomnia
Acronym: AURICULO-DODO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018_0107
Record Dates: First submitted 2020-06-10; First posted 2020-07-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Insomnia
Keywords: Cryo auriculotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryo-Auriculotherapy (Experimental): Patients benefit from 3 sessions of cryo-auriculotherapy with device with nitrous oxyde on 10 auricular points at one month intervals.
  Interventions: Device: Cryo-Auriculotherapy
- Control group (Sham Comparator): Patients benefit from 3 sessions of cryo-auriculotherapy with device without nitrous oxyde on 10 auricular points at one month intervals.
  Interventions: Device: Sham comparator

INTERVENTIONS:
Device: Cryo-Auriculotherapy — 3 sessions of cryo-auriculotherapy with device with nitrous oxyde on 10 auricular points at one month intervals.
  Arms: Cryo-Auriculotherapy
Device: Sham comparator — 3 sessions of cryo-auriculotherapy with device without nitrous oxyde on 10 auricular points at one month intervals.
  Arms: Control group

SUMMARY:
The aim of the study is to show that auriculotherapy is effective in the treatment of chronic insomnia.

DETAILED DESCRIPTION:
Chronic insomnia affects a significant proportion of the French population with an estimated prevalence between 15% and 20%.

This disease is mainly managed by general practitioners for whom benzodiazepines and Z-drugs (zopiclone, zolpidem) represent the first-line treatment. The french health authorities recommend limiting the consumption of these molecules to 2 to 4 weeks taking into account their possible undesirable effects (eg memory impairment, in the elderly, road accident) as well as the risk of tolerance and addiction. However, it appears that a majority of the patients concerned become chronic consumers.

The investigators propose to assess cryo-auriculotherapy in the treatment of chronic insomnia.

The population studied will consist of patients with chronic insomnia, whose diagnosis has been made according to the definition in the diagnostic and statistical manual of mental disorders (DSM-5), and followed up in an outpatient clinic at Foch Hospital or in one of the participating centers.

Half of the patients will be treated with cryo-auriculotherapy (use of a device with nitrous oxide) and compared with control patients who will have the same treatment visits involving a sham device (device without nitrous oxide).

ELIGIBILITY:
Inclusion Criteria:

* Suffering from chronic insomnia as defined in the diagnostic and statistical manual of mental disorders (DSM-5)
* Score ≥ 15 on the Insomnia Severity Index (ISI) questionnaire;
* Covered by a national healthcare insurance
* Consent form signed

Exclusion Criteria:

* Pregnant woman or pregnancy planned for the duration of the study;
* Regular night work or shift work / reversal of sleep patterns;
* Trans meridian travel during the previous month or planned during the study period;
* Unstable or untreated psychiatric disorder including severe depression, severe addiction, unbalanced bipolar disorder;
* Taking insomnia-inducing drugs (eg Corticoids);
* Hypnotic treatment or antidepressant treatment with hypnotic aim introduced since less than 4 weeks or with change dating back less than 4 weeks;
* Presence of organic comorbidities which may be responsible for sleep disorders (SAS and restless legs syndrome): (STOP-BANG) score ≥ 5;
* History of central neurological disorders or progressive brain injury;
* Contraindication to the use of auriculotherapy (lesion or infection of the pinna) by cryotherapy (skin scarring disorder, risk of hypo or hyperpigmentation);
* Treatment by auriculotherapy or acupuncture in this indication in the previous 12 months;
* Previous treatment with cryo-auriculotherapy
* Having started in the month preceding the first auriculotherapy session, any new treatment likely to interfere with the study: specific drug treatment (antidepressant, morphine or anticonvulsant) or complementary therapy (psychological care, physiotherapy, balneotherapy, etc.).
* Difficulty complying with the treatment, questionnaire or study protocol.
* Be deprived of liberty or under guardianship.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement of insomnia after 3 month of treatment (Real Auriculotherapy group compared to Sham Auriculotherapy group) | 3 months
  Comparison of the evolution of the score of the Insomnia Severity Index (7-item self-report questionnaire assessing the nature, severity, and impact of insomnia).
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
  The improvement will be defined as a decrease in the score of the questionnaire by 3 points between Day 90 and Day 0.
  A comparison of the improvement according to the 2 arms will be made.

SECONDARY OUTCOMES:
Evolution of sleep quality and sleep disorders | 3 months
  Specific questionnaire Pittsburgh Sleep Quality Index (PSQI)at inclusion and at 3 months (1 month post-treatment).
  Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21).
  Higher scores indicate worse sleep quality.
Evolution of drug consumption linked to chronic insomnia | 3 months
  Drugs used to control chronic insomnia will be collected from the inclusion to 3 months (1 month post-treatment)
Evolution and Anxiety and depression | 3 months
  Hospital Anxiety and Depression questionnaire will be used at inclusion and at 3 months post-treatment.
  There are seven questions related to anxiety (total A) and seven others related to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21).
  Higher score indicates a certain symptomatology :
  * 7 or less: absence of symptoms
  * 8 to 10: doubtful symptomatology
  * 11 and more: certain symptomatology.
Evolution of quality of life | 3 months
  EuroQoL five Dimension questionnaire at inclusion and at 3 months post-treatment. This questionnaire is designed for the patient to judge the impact of his state of health on his quality of life according to 5 dimensions (mobility, personal autonomy, daily activities, pain / discomfort and anxiety / depression). Each item has 3 response levels (1, 2 and 3) and the combination of the five digits will represent the patient's state of health. It is supplemented by a quality of life thermometer graduated from 0 (worst quality of life) to 100 (best quality of life).
Overall patient impression | 3 months
  Patient Global Impression of Change questionnaire (PGIC) used at the end of the follow-up.
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status with a seven-point single-item scale ranging from 'very much worse' to 'very much improved'
Willingness of the patient to continue treatment | 3 months
  Patient will be asked at the end of the study if they want to pursue the treatment
Tolerance of cryotherapy auriculotherapy treatment. | 3 months
  The presence or absence of adverse events attributed to the treatment of auriculotherapy by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - Espace Santé Simone Veil, Issy-les-Moulineaux, Hauts de Seine
  - Cabinet Médical Nouvelle France, Le Chesnay, Yvelines
  - Cabinet de l'Olivier, Montigny-le-Bretonneux, Yvelines
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No